CLINICAL TRIAL: NCT01730495
Title: Tumor Necrosis Factor-alpha Inhibition Using Etanercept in Moderate and Serious Chronic Fatigue Syndrome/ Myalgic Encephalomyelitis (CFS/ME), Including in Patients With no Clinical Response After B-lymphocyte Depletion Using the Anti-CD20 Antibody Rituximab.
Brief Title: Tumor Necrosis Factor-alpha Inhibition Using Etanercept in Chronic Fatigue Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: After inclusion of four patients, two experienced moderate worsening of symptoms
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011/2500; 2011-006069-16 (EudraCT Number)
Record Dates: First submitted 2012-11-08; First posted 2012-11-21 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Chronic Fatigue Syndrome; Myalgic Encephalomyelitis
Keywords: Chronic fatigue syndrome; CFS; Myalgic Encephalomyelitis (ME); CFS/ME; Tumor necrosis factor-alpha; TNF-alpha; Etanercept
MeSH Terms: conditions — Fatigue Syndrome, Chronic | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Etanercept (Experimental)
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — Weekly subcutaneous injections of Etanercept 50 mg, for up to 12 months.

SUMMARY:
The hypothesis is that a subset of patients with chronic fatigue syndrome/ myalgic encephalomyelitis (CFS/ME), including also patients with no clinical response after B-cell depletion therapy using the anti-CD20 antibody Rituximab, may benefit from tumor necrosis factor-alpha inhibition using Etanercept as weekly subcutaneous injections.

ELIGIBILITY:
Inclusion Criteria:

* chronic fatigue syndrome/ myalgic encephalomyelitis (CFS/ME)
* moderate and serious CFS/ME severity
* age 18-66 years
* informed consent

Exclusion Criteria:

* patients with fatigue, not fulfilling criteria for CFS
* pregnancy or lactation
* previous malignant disease, except basal cell carcinoma of skin and cervical carcinoma in situ
* previous long-term systemic treatment with immunosuppressive drugs such as cyclosporine, azathioprin, mycophenolate mofetil, except steroids e.g. in obstructive lunge disease.
* demyelinating disease, such as multiple sclerosis.
* heart failure.
* endogenous depression.
* lack of ability to comply to the protocol.
* multi-allergy with risk of serious drug reaction
* reduced renal function (creatinine > 1.5 x UNL)
* reduced liver function (bilirubin or transaminases > 1.5 x UNL)
* HIV positivity. Evidence of clinically significant infection. Previous viral hepatitis with risk of reactivation. High risk of opportunistic infections. Latent tuberculosis must be treated before inclusion.

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-10; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Symptom alleviation within 12 months follow-up, as compared to baseline, measured by standardized self-reports and quality of life schemes. | Response of at least six weeks duration, independent on when occuring, during 12 months follow-up.
  The primary endpoint is defined as moderate or major response of the CFS/ME symptoms, of at least six weeks duration, independent on when during 12 months follow-up the response period(s) occurs. Single such response periods, and the sum of these, are recorded.

SECONDARY OUTCOMES:
Symptom alleviation, as compared to baseline, measured by standardized self-reports and quality of life schemes. | At 3, 6, 9, 12 months after start of intervention.
  The secondary outcome measures are effect on the CFS/ME symptoms, by evaluation at 3, 6, 9, 12 months after start of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Øystein Fluge, MD, PhD, Principal Investigator — Dept. of Oncology and Medical Physics, Haukeland University Hospital
Locations (1):
- Dept. of Oncology and Medical Physics, Haukeland University Hospital Bergen, Norway, Bergen, Norway

REFERENCES:
- [Background] Fluge O, Bruland O, Risa K, Storstein A, Kristoffersen EK, Sapkota D, Naess H, Dahl O, Nyland H, Mella O. Benefit from B-lymphocyte depletion using the anti-CD20 antibody rituximab in chronic fatigue syndrome. A double-blind and placebo-controlled study. PLoS One. 2011;6(10):e26358. doi: 10.1371/journal.pone.0026358. Epub 2011 Oct 19. PMID 22039471
- [Background] Fluge O, Mella O. Clinical impact of B-cell depletion with the anti-CD20 antibody rituximab in chronic fatigue syndrome: a preliminary case series. BMC Neurol. 2009 Jul 1;9:28. doi: 10.1186/1471-2377-9-28. PMID 19566965